CLINICAL TRIAL: NCT00900614
Title: An Open-label Phase I Dose Escalating Study of APR-246 for Infusion in Patients With Refractory Hematologic Malignancies or Prostate Carcinoma
Brief Title: Safety Study of APR-246 in Patients With Refractory Hematologic Cancer or Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aprea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APR-246-01
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Hematologic Neoplasms; Prostatic Neoplasms
Keywords: Hematologic malignancy; Prostate carcinoma; Hematologic cancer; Prostate cancer
MeSH Terms: conditions — Hematologic Neoplasms; Prostatic Neoplasms | interventions — eprenetapopt

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: APR-246 — Intravenous infusion. Dose escalating. Dosing will be conducted with three patients at each dose level.

SUMMARY:
The purpose of this study is to determine the highest feasible dose (HFD) of intravenous (IV) APR-246 when given to patients with refractory hematologic malignancies or prostate carcinoma.

ELIGIBILITY:
Summary criteria for participant selection:

Inclusion Criteria:

* Male or female ≥ 18 years of age.
* Any below mentioned advanced disease, which is not eligible for other therapies. The diagnosis should have been confirmed either histologically or cytologically:

  1. Acute myeloid leukemia.
  2. Acute lymphoid leukemia.
  3. Chronic lymphocytic leukemia.
  4. Chronic myeloid leukemia.
  5. Chronic myelomonocytic leukemia.
  6. Multiple myeloma.
  7. Non Hodgkin's lymphoma.
  8. Hodgkin's lymphoma.
  9. Myelodysplastic syndrome.
  10. Myelofibrosis.
  11. Hormone refractory, metastatic prostate carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) is reached and HFD is defined accordingly, OR the dose, which is expected to result in maximum plasma concentration close to, but not exceeding 35 μg/ml in any single patient without showing signs of DLT. | 21 days

SECONDARY OUTCOMES:
Determination of the toxicity and safety profile of APR-246 based on safety parameters from the entire study period. | continuously during 21 days
Determination of the PK profile for up to 22 hours after the last APR-246 infusion. Cmax (maximal plasma concentration), AUC (area under the curve), t1/2 (half-life) and clearance will be determined. | continuously, during 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Sören Lehmann, MD, PhD, Principal Investigator — Hematology Centre, M54, Karolinska Institute, Karolinska University Hospital, Huddinge, SE-141 86, Stockholm, Sweden
Locations (6):
- Sweden (6):
  - Section of Haematology and Coagulation, Sahlgrenska University Hospital, Gothenburg
  - Department of Hematology, University Hospital, Örebro
  - Urology clinic, University Hospital, Örebro
  - Hematology Centre, M54, Karolinska Institute, Karolinska University Hospital, Huddinge, Stockholm
  - Clinical Research and Development Unit, Department of Oncology, Akademiska Hospital, Uppsala
  - Department of Haematology, Akademiska Hospital, Uppsala